CLINICAL TRIAL: NCT07340190
Title: A Phase 1b, Open Label, 2-Part Study to Evaluate the Effect of Pelabresib (DAK539/CPI-0610) on the Pharmacokinetics of Repaglinide, Midazolam, and Combined Drospirenone/Ethinyl Estradiol Oral Contraceptive in Patients With Advanced Malignancies
Brief Title: A Drug-drug Interaction Study to Evaluate the Effects of Pelabresib on the Pharmacokinetics of Repaglinide, Midazolam, and Combined Oral Contraceptive in Patients With Advanced Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDAK539A12102; 2025-521000-22-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignancies
Keywords: Drug-drug interaction (DDI); Cytochrome P450 (CYP); Advanced Malignancies; oral contraceptive; Pharmacokinetics (PK)
MeSH Terms: interventions — repaglinide; Midazolam; drospirenone; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Part 1 (PK profiles of victim drugs):
  • Arm A: repaglinide + midazolam + pelabresib
  Part 2 (Continued treatment):
  After completing Part 1, in case of clinical benefit, participants can continue with pelabresib treatment in Part 2 until the end of study (EOS) is reached or until the participant meets discontinuation criteria, or until they receive pelabresib treatment via alternative means of access, whichever occurs first.
  Interventions: Drug: pelabresib; Drug: repaglinide; Drug: midazolam
- Arm B (Experimental): Part 1 (PK profiles of victim drugs):
  • Arm B: drospirenone + ethinyl estradiol + pelabresib
  Part 2 (Continued treatment):
  After completing Part 1, in case of clinical benefit, participants can continue with pelabresib treatment in Part 2 until the end of study (EOS) is reached or until the participant meets discontinuation criteria, or until they receive pelabresib treatment via alternative means of access, whichever occurs first.
  Interventions: Drug: pelabresib; Drug: drospirenone; Drug: ethinyl estradiol

INTERVENTIONS:
Drug: pelabresib — pelabresib 225 mg orally (PO) once daily (QD) for 14 days, followed by a 7-day break
  Other Names: DAK539 (formerly CPI-0610)
Drug: repaglinide — 0.5 mg repaglinide tablet administered orally on Pre-Cycle Day 1 and Cycle 1 Day 14
  Arms: Arm A
Drug: midazolam — 2 mg/mL midazolam oral solution administered orally on Pre-Cycle Day 1 and Cycle 1 Day 14
  Arms: Arm A
Drug: drospirenone — 3 mg drospirenone tablet administered orally on Pre-Cycle Day 1 and Cycle 1 Day 10
  Arms: Arm B
Drug: ethinyl estradiol — 0.03 mg ethinyl estradiol tablet administered orally on Pre-Cycle Day 1 and Cycle 1 Day 10
  Arms: Arm B

SUMMARY:
This drug-drug interaction (DDI) study aims to evaluate the impact of pelabresib at steady-state plasma concentrations on the pharmacokinetic (PK) profile of A) a single dose of repaglinide and a single dose of midazolam, and B) a single dose of combined drospirenone and ethinyl estradiol. The study will be conducted in adult participants with advanced malignancies for whom no standard or curative treatment options are available.

DETAILED DESCRIPTION:
This clinical study is divided into two components:

1. Part 1: Interventional Phase This phase evaluates the drug-drug interaction (DDI) potential of pelabresib with specific victim drugs.

   * Arm A: Assesses pelabresib's DDI potential with repaglinide and midazolam. Participants will be hospitalized for two nights-one starting on Pre-cycle Day 1 and another on Day 14. Beginning Cycle 1 Day 1, participants will receive 225 mg of pelabresib daily for 14 days, followed by a 7-day break.
   * Arm B: Evaluates pelabresib's DDI potential with drospirenone and ethinyl estradiol. Hospitalization will range from a minimum of 2 nights to a maximum of 10 nights-up to 5 nights starting on Pre-cycle Day 1, and up to 5 nights starting on Cycle 1 Day 10. Participants will follow the same pelabresib dosing schedule as Arm A. Arm B will proceed independently of Arm A's results.
2. Part 2: Continued Treatment Phase Participants demonstrating clinical benefit, as determined by the investigator, may continue receiving pelabresib in additional treatment cycles.

A participant is considered to have entered the screening period upon signing the informed consent form. Enrollment occurs when the participant is assigned their first dose of study treatment via the IRT system. Completion is defined as having finished all study phases, including the End of Treatment (EOT) and the 30-day Safety Follow-Up visits. Participants with hematological malignancies will continue follow-up every 3 months after EOT.

1. End of Treatment Visit Must occur within 7 days of the last pelabresib dose or within 7 days of the decision to discontinue treatment, if that decision is made more than 7 days after the last dose.
2. 30-Day Safety Follow-Up All participants will be monitored for adverse events (AEs) and serious adverse events (SAEs) for 30 ± 3 days after the final pelabresib dose. If a participant initiates another anticancer therapy or transitions to pelabresib via another source (e.g., extension study or commercial supply), safety follow-up ends at the start of the new treatment.
3. Leukemic Transformation Monitoring Participants with hematological malignancies will be followed every 3 months after EOT for signs of leukemic transformation, continuing until one of the following: study end, confirmation of acute myeloid leukemia (AML), withdrawal of consent, loss to follow-up, or death.

ELIGIBILITY:
Key Inclusion Criteria:

Key inclusion criteria for all participants (Arm A and Arm B)

* Is at least 18 years of age at the time of signing the informed consent.
* Has a confirmed documented diagnosis of an advanced malignancy for which no standard and/or curative treatment options are available
* Has the following acceptable laboratory assessments prior to the first dose of study treatment:

  1. Platelet count ≥ 150 × 109 /L in the absence of thrombopoietic factors or transfusions within 2 weeks of the screening assessment
  2. Absolute neutrophil count (ANC) ≥ 1 × 109 /L in the absence of granulocyte growth factors
  3. Peripheral blood blast count < 5%. Assessment of blasts in bone marrow is not mandatory at screening; however, blasts must be <5% if the bone marrow assessment is performed.
  4. Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN)
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN (≤5 × ULN if the elevation can be ascribed to liver involvement)
  6. Calculated or measured creatinine clearance of ≥30 mL/min*
* Has fully recovered from major surgery and from the acute toxic effects of prior chemotherapy and radiotherapy (residual Grade 1 toxicities and residual alopecia of any grade are allowed).

Additional inclusion criterion for Arm B

• Is a female participant.

Key Exclusion Criteria:

Key exclusion criteria for Arm A

* Has a history of hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical class.
* Is pregnant (confirmed by a pregnancy test at screening) or is breastfeeding.
* Has current known active or chronic infection with HIV, hepatitis B, or hepatitis C.
* Has impaired cardiac function or clinically significant cardiac disease.
* Has a gastrointestinal tumor, impaired GI function, GI disease, or significant resection of stomach or other portion of the gastrointestinal tract that could alter the absorption of pelabresib, midazolam, or repaglinide, including any unresolved nausea, vomiting, or diarrhea.

Key exclusion criteria for Arm B

* Has renal impairment (CrCl less than 50 mL/min).
* Has a gastrointestinal tumor, impaired GI function, GI disease, or significant resection of stomach or other portion of the gastrointestinal tract that could alter the absorption of pelabresib, drospirenone and ethinyl estradiol, including any unresolved nausea, vomiting, or diarrhea.
* Has breast cancer or other estrogen- or progestin-sensitive cancer.
* Has undiagnosed abnormal uterine bleeding.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-05-29 (Estimated); Primary Completion 2029-11-15 (Estimated); Study Completion 2029-12-14 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of repaglinide, midazolam, and drospirenone and ethinyl estradiol | Arm A: Pre-Cycle Day 1/Cycle 1 Day 14 (Predose, 0.25-12 hours); Cycle 1 Days 1/15 (24 hours). Arm B: Pre-Cycle Day 1/Cycle 1 Day 10 (Predose, 0.5-10 hours); Days 2/11 (24 h), 3/12 (48 h), 4/13 (72 h), 5/14 (96 h); Cycle 1 Days 1/15 (120 h). 21-day cycle.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax of repaglinide, midazolam and combined oral contraceptive drospirenone and ethinyl estradiol per study group will be listed and summarized using descriptive statistics
Time to Maximum Concentration (Tmax) of repaglinide, midazolam, and drospirenone and ethinyl estradiol | Arm A: Pre-Cycle Day 1/Cycle 1 Day 14 (Predose, 0.25-12 hours); Cycle 1 Days 1/15 (24 hours). Arm B: Pre-Cycle Day 1/Cycle 1 Day 10 (Predose, 0.5-10 hours); Days 2/11 (24 h), 3/12 (48 h), 4/13 (72 h), 5/14 (96 h); Cycle 1 Days 1/15 (120 h). 21-day cycle.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax of repaglinide, midazolam and combined oral contraceptive drospirenone and ethinyl estradiol per study group will be listed and summarized using descriptive statistics
Area Under the Curve to Last Measurable Concentration (AUClast) of repaglinide, midazolam, and drospirenone and ethinyl estradiol | Arm A: Pre-Cycle Day 1/Cycle 1 Day 14 (Predose, 0.25-12 hours); Cycle 1 Days 1/15 (24 hours). Arm B: Pre-Cycle Day 1/Cycle 1 Day 10 (Predose, 0.5-10 hours); Days 2/11 (24 h), 3/12 (48 h), 4/13 (72 h), 5/14 (96 h); Cycle 1 Days 1/15 (120 h). 21-day cycle.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast of repaglinide, midazolam and combined oral contraceptive drospirenone and ethinyl estradiol per study group will be listed and summarized using descriptive statistics
Area Under the Curve to Infinity (AUCinf) of repaglinide, midazolam, and drospirenone and ethinyl estradiol | Arm A: Pre-Cycle Day 1/Cycle 1 Day 14 (Predose, 0.25-12 hours); Cycle 1 Days 1/15 (24 hours). Arm B: Pre-Cycle Day 1/Cycle 1 Day 10 (Predose, 0.5-10 hours); Days 2/11 (24 h), 3/12 (48 h), 4/13 (72 h), 5/14 (96 h); Cycle 1 Days 1/15 (120 h). 21-day cycle.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUCinf of repaglinide, midazolam and combined oral contraceptive drospirenone and ethinyl estradiol per study group will be listed and summarized using descriptive statistics

SECONDARY OUTCOMES:
Apparent Clearance (CL/F) of repaglinide, midazolam, and drospirenone and ethinyl estradiol | Arm A: Pre-Cycle Day 1/Cycle 1 Day 14 (Predose, 0.25-12 hours); Cycle 1 Days 1/15 (24 hours). Arm B: Pre-Cycle Day 1/Cycle 1 Day 10 (Predose, 0.5-10 hours); Days 2/11 (24 h), 3/12 (48 h), 4/13 (72 h), 5/14 (96 h); Cycle 1 Days 1/15 (120 h). 21-day cycle.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL/F of repaglinide, midazolam and combined oral contraceptive drospirenone and ethinyl estradiol per study group will be listed and summarized using descriptive statistics.
Apparent Volume of Distribution during Terminal Phase (Vz/F) of repaglinide, midazolam, and drospirenone and ethinyl estradiol | Arm A: Pre-Cycle Day 1/Cycle 1 Day 14 (Predose, 0.25-12 hours); Cycle 1 Days 1/15 (24 hours). Arm B: Pre-Cycle Day 1/Cycle 1 Day 10 (Predose, 0.5-10 hours); Days 2/11 (24 h), 3/12 (48 h), 4/13 (72 h), 5/14 (96 h); Cycle 1 Days 1/15 (120 h). 21-day cycle.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz/F of repaglinide, midazolam and combined oral contraceptive drospirenone and ethinyl estradiol per study group will be listed and summarized using descriptive statistics.
Terminal Half-Life (T½) of repaglinide, midazolam, and drospirenone and ethinyl estradiol | Arm A: Pre-Cycle Day 1/Cycle 1 Day 14 (Predose, 0.25-12 hours); Cycle 1 Days 1/15 (24 hours). Arm B: Pre-Cycle Day 1/Cycle 1 Day 10 (Predose, 0.5-10 hours); Days 2/11 (24 h), 3/12 (48 h), 4/13 (72 h), 5/14 (96 h); Cycle 1 Days 1/15 (120 h). 21-day cycle.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. T½ of repaglinide, midazolam and combined oral contraceptive drospirenone and ethinyl estradiol per study group will be listed and summarized using descriptive statistics
Maximum Plasma Concentration (Cmax) of pelabresib at steady state | Arm A: Pre-Cycle Day 1/Cycle 1 Day 14 (Predose, 0.25-12 hours); Cycle 1 Days 1/15 (24 hours). Arm B: Pre-Cycle Day 1/Cycle 1 Day 10 (Predose, 0.5-10 hours); Days 2/11 (24 h), 3/12 (48 h), 4/13 (72 h), 5/14 (96 h); Cycle 1 Days 1/15 (120 h). 21-day cycle.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax of pelabresib at steady state per study group will be listed and summarized using descriptive statistics.
Area Under the Curve from 0 to 24 hours on Day 14 (AUC₀-24h) of pelabresib at steady state | Arm A: Pre-Cycle Day 1/Cycle 1 Day 14 (Predose, 0.25-12 hours); Cycle 1 Days 1/15 (24 hours). Arm B: Pre-Cycle Day 1/Cycle 1 Day 10 (Predose, 0.5-10 hours); Days 2/11 (24 h), 3/12 (48 h), 4/13 (72 h), 5/14 (96 h); Cycle 1 Days 1/15 (120 h). 21-day cycle.
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC₀-24h of pelabresib at steady state per study group will be listed and summarized using descriptive statistics.
Number of Participants with adverse events (AEs), serious AEs (SAEs) | Through study completion, an average of 42 months
  Incidence of adverse events by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No